CLINICAL TRIAL: NCT07388030
Title: Lithotripsy Versus Balloon Angioplasty for Optimal Treatment of CAlcified Lesions With and Without Optical Coherence Tomography evaluatION
Acronym: LOCATION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Bluesail Boyuan Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LFBY-202504
Record Dates: First submitted 2026-01-15; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: CAD - Coronary Artery Disease; Severe Coronary Calcified Lesions
Keywords: severe coronary calcified lesions; intravascular lithotripsy (IVL); balloon angioplasty (BA); optical coherence tomography (OCT)-guided; angiography-guided; target vessel failure (TVF); percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: The LOCATION study adopts a **prospective, multicenter, 2×2 factorial randomized controlled model** for severe coronary calcified lesions.
  Key details:
  1. **Randomization**: 3,060 patients are 1:1 randomized to IVL/BA pretreatment and 1:1 to OCT/angiography guidance (4 parallel groups), stratified by site and diabetes with block sizes 2/4/6 via IWRS.
  2. **Interventions**: IVL (SoniCracker™) vs standard BA for lesion prep; OCT (Nanjing Forssmann) vs angiography for stent guidance.
  3. **Crossover Rules**: BA→IVL prohibited; IVL→other devices allowed only for specific criteria (recorded as failure).
  4. **Blinding**: Open-label for investigators/subjects; core lab and CEC adjudicate outcomes blindly.
  5. **Follow-up**: 30 days, 6 months, 1/2/3 years + sweep visit; primary endpoint is 3-year TVF.
  6. **Analysis Sets**: ITT (efficacy), PP (sensitivity), SS (safety).
Who Masked: Outcomes Assessor
Masking Description: In addition to the Outcomes Assessor, the following parties are also masked in the clinical trial:
  Imaging Core Laboratory Personnel: They perform blinded quantitative analysis on all baseline and post-procedural coronary angiography images, as well as blinded analysis on final OCT images. They are unaware of the subjects' randomized treatment groups to ensure the objectivity of imaging evaluation results.
  Clinical Events Committee (CEC) Members: They conduct blinded adjudication of primary and secondary endpoint events (such as target vessel failure, myocardial infarction, etc.). Without knowing the subjects' treatment assignments, they assess the occurrence and severity of events to avoid bias in endpoint judgment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IVL pre-treatment plus OCT-guided group (Experimental): (1st OCT) perform OCT after the small balloon pre-dilatation but before the IVL; then IVL is performed* followed by the 1:1 high-pressure balloon pre-dilatation followed by the 2nd OCT; then implant the DES and perform post-dilatation with a high-pressure balloon at ≥18 atm (mandatory); then perform the final OCT (3rd OCT). Assess the stent to determine if further PCI is required to optimize stent implantation - either maximize stent expansion or treat malapposition, tissue protrusion, a major edge dissection or untreated reference segment disease. If further stent optimization is required, do so, after which a final OCT run must be performed again (4th OCT). Note: If IVL is unable to cross or dilate the lesion, rotational atherectomy, orbital atherectomy, or excimer laser should be performed followed by IVL. OCT must still be performed prior to stenting. Investigators should use IVL in accordance with the device's instructions for use.
  Interventions: Device: IVL Pretreatment + OCT-Guided Stent Implantation
- IVL pre-treatment plus angiography-guided group (Active Comparator): An attempt should be made to cross the target lesion with the IVL catheter after the 1.5 mm or 2.0 mm balloon dilation. If the IVL will not cross the lesion, a larger balloon or atherectomy may be used - then IVL must be performed*. Following successful IVL, pre-dilatation must be performed and be successful (complete balloon expansion) with a high-pressure balloon sized 1:1 to the distal reference segment prior to stenting (mandatory); then one or more stents are implanted (DES only); then post-dilatation must be performed with a high-pressure balloon at ≥18 atm (mandatory). A final OCT run blinded to the operator is then performed as the last procedure. NOTE: Investigators should use IVL in accordance with the device's instructions for use.
  Interventions: Device: IVL Pretreatment + Angiography-Guided Stent Implantation
- balloon angioplasty pre-treatment plus OCT-guided group (Active Comparator): (1st OCT) perform baseline OCT after the 1.5 or 2.0 mm balloon; then perform balloon pre-dilatation with a high-pressure balloon sized 1:1 to the distal RVD*; then perform OCT again (2nd OCT); then implant the DES and perform post-dilatation with a high-pressure balloon at ≥18 atm (mandatory); then perform the final OCT (3rd OCT). Assess the stent to determine if further PCI is required to optimize stent implantation - either maximize stent expansion or treat malapposition, tissue protrusion, a major edge dissection or untreated reference segment disease. If further stent optimization is required, do so, after which a final OCT run must be performed again (4th OCT).
  Interventions: Device: Balloon Angioplasty (BA) Pretreatment + OCT-Guided Stent Implantation
- balloon angioplasty pre-treatment plus angiography-guided group (Active Comparator): pre-dilatation must be successful (complete balloon expansion) with a high-pressure balloon (or scoring balloon, cutting balloon, etc.) sized 1:1 to the distal reference segment (mandatory)*; then one or more stents are implanted (DES only); then post-dilatation must be performed with a high-pressure balloon at ≥18 atm (mandatory). *Note: if the 1:1 pre-dilatation balloon is unable to be fully expanded, rotational atherectomy, orbital atherectomy, or excimer laser may be performed. Crossover to IVL is not allowed. After atherectomy or excimer laser, the lesion must again be successfully pre-dilated (complete balloon expansion) with a high-pressure balloon sized 1:1 to the distal reference segment (mandatory) prior to stenting. A final OCT run blinded to the operator is then performed as the last procedure;
  Interventions: Device: Balloon Angioplasty (BA) Pretreatment + Angiography-Guided Stent Implantation

INTERVENTIONS:
Device: IVL Pretreatment + OCT-Guided Stent Implantation — Subjects who have signed ICF and have met all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 to IVL vessel preparation strategy or balloon angioplasty vessel preparation strategy. Concurrently, subjects will randomly be assigned in a 1:1 ratio to receive OCT-guidance or angiographic-guidance of the PCI procedure.
  Subject randomization in each of the 4 groups will be stratified by site and diabetes in varying block sizes of 2, 4 or 6. Randomization will be conducted with the use of an interactive web response system (IWRS).
  Arms: IVL pre-treatment plus OCT-guided group
Device: IVL Pretreatment + Angiography-Guided Stent Implantation — Subjects who have signed ICF and have met all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 to IVL vessel preparation strategy or balloon angioplasty vessel preparation strategy. Concurrently, subjects will randomly be assigned in a 1:1 ratio to receive OCT-guidance or angiographic-guidance of the PCI procedure.
  Subject randomization in each of the 4 groups will be stratified by site and diabetes in varying block sizes of 2, 4 or 6. Randomization will be conducted with the use of an interactive web response system (IWRS).
  Arms: IVL pre-treatment plus angiography-guided group
Device: Balloon Angioplasty (BA) Pretreatment + OCT-Guided Stent Implantation — Subjects who have signed ICF and have met all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 to IVL vessel preparation strategy or balloon angioplasty vessel preparation strategy. Concurrently, subjects will randomly be assigned in a 1:1 ratio to receive OCT-guidance or angiographic-guidance of the PCI procedure.
  Subject randomization in each of the 4 groups will be stratified by site and diabetes in varying block sizes of 2, 4 or 6. Randomization will be conducted with the use of an interactive web response system (IWRS).
  Arms: balloon angioplasty pre-treatment plus OCT-guided group
Device: Balloon Angioplasty (BA) Pretreatment + Angiography-Guided Stent Implantation — Subjects who have signed ICF and have met all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 to IVL vessel preparation strategy or balloon angioplasty vessel preparation strategy. Concurrently, subjects will randomly be assigned in a 1:1 ratio to receive OCT-guidance or angiographic-guidance of the PCI procedure.
  Subject randomization in each of the 4 groups will be stratified by site and diabetes in varying block sizes of 2, 4 or 6. Randomization will be conducted with the use of an interactive web response system (IWRS).
  Arms: balloon angioplasty pre-treatment plus angiography-guided group

SUMMARY:
Severely calcified coronary artery disease means that calcium has built up in the blood vessels that supply the heart. This makes coronary procedures more difficult and increases the risk of complications during and after treatment.

The LOCATION Study is a large clinical study designed to compare different commonly used treatment strategies for patients with severely calcified coronary arteries who need a coronary stent. The study aims to find safer and more effective ways to prepare the artery and place the stent in order to improve long-term outcomes.

In this study, participants will be randomly assigned (like flipping a coin) to one of four treatment groups during their coronary procedure. The treatments differ in two ways: (1) how the calcified artery is prepared before placing the stent, and (2) how imaging is used to guide stent placement.

One method uses a shockwave-based device to help break calcium in the artery, while the other uses standard balloon treatment. For imaging guidance, one approach uses a high-resolution imaging catheter inside the artery, and the other relies on standard X-ray imaging. All participants will receive a standard, approved drug-eluting stent as part of routine care.

The main goal of the study is to determine which treatment approach best reduces serious heart-related problems over three years. These problems include heart-related death, heart attack in the treated vessel, or the need for another procedure on the same vessel.

Adults aged 18 years or older with significant coronary artery narrowing and severe calcium buildup may be eligible to participate. All participants must provide written informed consent before joining the study.

Participants will be followed during their hospital stay and through regular follow-up visits or phone calls for up to three years after the procedure. Information collected during the study will help doctors better understand how to treat patients with severely calcified coronary arteries in the future.

Participation in this study is voluntary, and patients may withdraw at any time without affecting their medical care. All study devices used in this trial are approved for clinical use, and patient privacy will be protected according to applicable regulations.

DETAILED DESCRIPTION:
LOCATION Study is a prospective, multicenter, 2x2 factorial randomized controlled trial.

Number of Sites: Approximately 50 sites in China.

Trial Objectives:

Objective 1: To evaluate the efficacy and safety of coronary intravascular lithotripsy (IVL) compared with balloon angioplasty (BA) for pretreatment of severely coronary calcified lesions prior to implantation of stents.

Objective 2: To evaluate the efficacy of optical coherence tomography (OCT)-guided compared with angiography-guided stent implantation in severely coronary calcified lesions.

Trial Hypotheses:

Hypotheses 1: IVL pretreatment of severely calcified coronary artery lesions will reduce the 3-year risk of target vessel failure (TVF, a composite of cardiac death, target vessel myocardial infarction [TVMI], or clinically-driven target vessel revascularization [TVR]) compared with BA pretreatment.

Hypotheses 2: OCT-guided percutaneous coronary intervention (PCI) will reduce 3-year risk of TVF compared with angiography-guided PCI in severely coronary calcified lesions.

Trial Population:Patients with one or more angiographically severely calcified coronary lesions

Trial Devices:

IVL device: SoniCrackerTM Coronary IVL Therapy System (Shanghai Bluesail Boyuan Medical Technology co., Ltd) BA Devices: standard commercially approved balloon angioplasty devices including high-pressure balloons, scoring balloons, and cutting balloons, without brand restriction OCT device: Intravascular Imaging System (Nanjing Forssmann Medical Technology Co., Ltd)

Follow-up Visits:

Follow-up will range between 1-year minimum and 3-year maximum. Follow-up will be conducted at discharge, at 30 (±7) days, 180 (±7) days, at 1 year (±30 days), 2 years (±30 days), at 3 (±30 days) years with clinic visit or phone calls. When the last patient reaches 1 year follow-up, an additional "sweep visit" will be performed in all patients who have not had follow-up within 30 days. Additional visits will not be performed after this sweep visit.

Duration:The period of this trial is expected to be approximately 4 years.

Sample size Calculation:

This trial is expected to enroll 3,060 patients, and the sample size calculation is based on the cumulative incidence of TVF as the primary endpoint.

For Hypothesis 1: We expect that the rate of TVF in the BA group will be 7.0%, 12.5%, 16.0% at 1-year, 2-year, and 3-year follow-up, respectively. Assuming a 25% risk reduction, (i.e. the hazard ratio (HR) between the IVL group and the BA group is 0.75), it is estimated that the rate of TVF in the IVL group will be 5.3%, 9.4%, and 12.0% at 1-year, 2-year, and 3-year follow-up, respectively. The subject enrollment period is expected to be 3 years, with annual enrollment rates of 30%, 40%, and 30% respectively. Accounting for a 5% dropout rate in both groups, 3,060 total randomized patients provide 80% power to reject the null hypothesis at a two-sided α level of 0.05.

For Hypothesis 2: We expected that the rate of TVF in the angiography-guided group will be 7.7%, 13.8%, 17.6% at 1-year, 2-year, and 3-year follow-up, respectively. Assuming a 27% risk reduction (i.e. the HR between the OCT-guided group and the angiography-guided group is 0.73), the rate of TVF in the OCT-guided group will be 5.6%, 10.1%, and 12.9% at 1-year, 2-year, and 3-year follow-up, respectively. The subject enrollment period is expected to be 3 years, with annual enrollment rates of 30%, 40%, and 30% respectively. Accounting for a 5% dropout rate in both groups, 2,326 total randomized patients provide 80% power to reject the null hypothesis at a two-sided α level of 0.05. With 3,060 total subjects, 89.6% power is present to reject the null hypothesis.

No interaction between hypotheses 1 and 2 are expected; that is, the benefit of OCT guidance is expected to accrue to a similar degree after both IVL and BA pre-treatment of severely calcified lesions; as such, adjustment for multiplicity is not required. Thus, a total enrollment of 3,060 subjects is planned, with 1530 subjects in each group (IVL vs. BA vessel preparation, and OCT vs. angiography guidance).

Background:

Coronary artery disease (CAD) is a major cardiovascular disorder that imposes a substantial burden on global health. Percutaneous coronary intervention (PCI), as an effective therapeutic strategy for CAD, has been increasingly utilized in clinical practice. With the aging of the population, the proportion and severity of coronary artery calcified lesions have shown a progressive increase. Severely calcified lesions represent one of the most prevalent complex lesion subtypes in CAD that significantly increases the technical difficulty of coronary intervention and thus poses a major challenge to cardiovascular interventional physicians. Notably, patients with calcified lesions have a significantly higher incidence of perioperative complications and long-term major adverse cardiovascular events (MACE). [1] For the pretreatment of calcified lesions, specialized balloons are typically employed, including high-pressure non-compliant balloons, cutting balloons and scoring balloons, as well as coronary atherectomy. However, these approaches have certain limitations. For instance, coronary atherectomy modifies lesion compliance and enlarges the lumen through the ablation of calcified plaques; yet, it may increase the risk of distal embolization, which can result in slow flow or no-reflow. Additionally, its complexity impedes its widespread adoption. Meanwhile, cutting balloons and scoring balloons have not been proven to enhance clinical outcomes in severe calcification.

Coronary intravascular lithotripsy (IVL) is derived from urological lithotripsy techniques. The IVL system consists of miniaturized, arrayed lithotripsy emitters enclosed within a balloon that generate a localized field effect at calcified sites, thereby optimizing energy delivery for the treatment of coronary calcification. This process modifies vascular compliance while preserving the integrity of the native fibroelastic components of the vessel wall, thus reducing vascular injury. The DISRUPT CAD I trial (NCT02650128) [2], the first study investigating IVL, enrolled 60 patients and demonstrated a 98% device success rate for IVL. Following IVL, all patients underwent successful drug-eluting stent (DES) implantation. Subsequently, a series of prospective, multicenter studies have been conducted, including DISRUPT CAD II (NCT03328949) [3], DISRUPT CAD III (NCT03595176) [4-5], and Disrupt CAD IV (NCT04151628) [6-7]. These studies have demonstrated the efficacy and safety of IVL in the management of severe coronary calcified lesions.

The SoniCrackerTM Coronary Intravascular Lithotripsy Therapy System is an IVL product developed by Shanghai Bluesail Boyuan Medical Technology co., Ltd. The device has completed a prospective, multicenter, single-arm pre-market clinical study, enrolling a total of 184 patients with severe coronary artery calcification in China, which showed a procedural success rate of 96.7% (defined as a residual in-stent stenosis ≤30% following stent implantation and without in-hospital major adverse cardiac events). Angiographic success (defined as residual in-stent stenosis ≤30% following stent implantation and without serious angiographic complications) and device success (defined as the IVL catheter successfully crossing the target lesion and delivering lithotripsy without serious angiographic complications) rates were both 100%, with no cases of post-stent residual stenosis >30% or severe angiographic complications. No intraoperative MACE occurred, and the postoperative 6-month MACE rate was 4.9%. The target lesion failure (TLF) rates at 1 month and 6 months post-procedure were 3.3% and 4.4%, respectively. Optical coherence tomography (OCT) subgroup analysis showed immediate post-procedure minimum stent area of 5.30±1.74 mm², minimum stent lumen diameter of 2.56±0.42 mm, immediate lumen gain diameter of 0.98±0.57 mm, and immediate lumen gain area of 3.29±1.45 mm² (data not published). The trial confirmed the device's favorable safety and efficacy. However, there is currently a lack of randomized controlled clinical trial data comparing IVL technology with other calcified lesion management strategies to further validate the superiority of IVL.

Current guidelines recommend the use of intravascular imaging guidance during PCI for complex coronary lesions (especially left main, true bifurcation, and long lesions). However, there remains a lack of intravascular imaging-guided studies with sufficient statistical power to confirm its efficacy in severely calcified lesions. Common clinical intravascular imaging modalities primarily include intravascular ultrasound (IVUS) and OCT. Compared to IVUS, OCT offers distinct advantages in evaluating calcified lesions: it can precisely assess calcification thickness and more accurately quantify the volume of calcified lesions, which is of great significance for determining optimal treatment strategies. Therefore, this trial is designed to evaluate the clinical benefits of OCT-guided stent implantation specifically in severe coronary calcified lesions.

The present clinical trial will employ the SoniCracker™ Coronary Intravascular Lithotripsy Therapy System and Intravascular Imaging System (Nanjing Forssmann Medical Technology Co., Ltd) to further evaluate two key aspects: first, the efficacy and safety of IVL using the SoniCracker™ system versus balloon angioplasty as pretreatment for severely coronary calcified lesions prior to stent implantation; second, the efficacy and safety of OCT-guided versus angiography-guided stent implantation in severely coronary calcified lesions.

Analysis of Potential Benefits

The devices used in the trial have demonstrated safety and efficacy in pre-market clinical trials and has obtained marketing approval from the China National Medical Products Administration (NMPA). Potential benefits include: achieving immediate procedural success, adequate stent expansion, reducing intraoperative complications, improving long-term vascular patency, and clinical outcomes, etc. Participation in this trial is purely voluntary, and enrolled subjects will not receive direct additional benefits. However, information collected from this trial may help deepen the understanding of clinical outcomes in percutaneous coronary intervention (PCI). Ultimately, this knowledge may provide physicians with more information to help improve the treatment of future patients.

Data Management System

The data collection/management system for this trial is an EDC (Electronic Data Capture) system. This is a validated electronic data capture system with audit trial management and user permission management capabilities.

Source data verification is performed to ensure the accuracy and completeness of key study variables. Protocol deviations, adverse events, and serious adverse events are documented and reported according to the study protocol and applicable regulatory and local regulatory requirements.

General Principles

Continuous variables will be summarized as the number of observations, number of missing values, mean, standard deviation, median, quartiles, and range. Categorical variables will be summarized as the number of observations, number of missing values, frequencies, and percentages. Baseline clinical, demographic, laboratory and procedural characteristics will be summarized by randomized treatment group.

All statistical analyses will be performed using SAS software, Version 9.4 or greater. For comparison between the two groups, all hypothesis tests are conducted by two-sided test, α=0.05. The efficacy analysis will be conducted according to the intention-to-treat (ITT) principle. Kaplan-Meier curves and log-rank test will be used to analyze and compare the timing of the first event in each group. P <0.05 is statistically significant. The reliability of all 2-sided confidence intervals (CI) is 95%, and Cox proportional risk regression model is used to determine the hazard ratio (HR).

Ethical Considerations

The study is conducted in compliance with the Declaration of Helsinki, applicable regulatory requirements, and approvals from institutional review boards or ethics committees at each participating site. All participants provide written informed consent prior to enrollment. Participant confidentiality is maintained throughout the study.

The Clinical Events Committee (CEC) will be established for this study.The Crossover Device Evaluation Committee will be established to provide impartial assessment of crossover subjects.The imaging core lab(s) will provide central reading/analysis for angiographic and OCT images generated pre-procedure,during the procedure, and post-procedure at enrolling sites.

Data Safety Monitoring Board (DSMB)

A Data Safety Monitoring Board will be established for this clinical trial to assess, at intervals during the trial, the data and to recommend to the Steering Committee whether to continue, suspend, modify, or terminate the trial early. The DSMB will consist of a minimum of three (3) members, one of which will be a statistician. The DSMB will not be affiliated with the Sponsor or its members will not be actively participating in the trial. Details of the DSMB's composition, specific review processes, and operating procedures are outlined in its charter.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion criteria:

  1. Age ≥18 years;
  2. Subject presents with:

     1. stable ischemic heart disease or
     2. acute coronary syndrome (non-ST-segment elevation myocardial infarction [NSTEMI] or unstable angina), or
     3. stabilized recent ST-segment elevation myocardial infarction (STEMI) (>48 hours prior to enrollment);
  3. Subject has been fully informed and signed the Institutional Review Board (IRB) approved LOCATION trial Informed Consent Form (ICF) prior to any trial related procedures.
* Angiographic inclusion criteria：

  1. The reference diameter of each target vessel is ≥2.25 mm and ≤4.0 mm at the lesion site (visual estimation);
  2. The target lesion(s) have:

  <!-- -->

  1. A stenosis ≥70% and <100% (visual estimation), or
  2. A stenosis of the target lesion ≥50% and <70% (visual estimation) with evidence of ischemia via:

     1. Positive stress testing (such as single-photon emission computed tomography, echocardiography, treadmill exercise test, etc.), or computed tomography-fractional flow reserve (CT-FFR) value ≤0.80, or;
     2. 24-hour Holter electrocardiogram: ST-segment elevation or depression of ≥1 mm in horizontal or down-sloping pattern lasting for at least 1 minute, with an interval of more than 1 minute between two episodes; combined with the patient presenting typical angina symptoms with Canadian Cardiovascular Society grading of angina pectoris II - IV;
     3. Pressure wire FFR or angioFFR value ≤0.80 or instantaneous wave-free ratio (iFR) value ≤0.89.

        3.The target lesion has fluoroscopic evidence of severe calcium at the lesion site, defined via angiogram as fluoroscopic radiopacities noted without cardiac motion before contrast injection involving both sides of the arterial wall in at least 1 location and total length of calcium of at least 15 mm; All lesions in the non-target vessel, if any, that require treatment are successfully treated without complications prior to randomization, defined as final diameter stenosis ≤20% with final TIMI-3 flow, with no residual dissection grade ≥type B, and no transient or sustained angiographic complications (e.g. distal embolization, side branch closure), no chest pain lasting >5 minutes, and no ST-segment elevation or depression lasting >5 minutes.

        Exclusion Criteria:
* Clinical exclusion criteria：

  1. Subject has undergone PCI in the target vessel or its branches within 12 months prior to randomization or prior CABG any time;
  2. Subject has undergone a PCI procedure in a non-target vessel that is unsuccessful or with complications within 30 days prior to randomization, including during the randomization procedure. Successful and uncomplicated PCI is defined as final diameter stenosis ≤20% with final TIMI-3 flow, no residual dissection grade≥ type B, no transient or sustained angiographic complications (e.g., distal embolization, side branch closure), no chest pain lasting >5 minutes, and no ST-segment elevation or depression lasting >5 minutes);
  3. PCI is planned within 12 months post randomization aside from a potential planned staged PCI as part of the randomized treatment strategy;
  4. Planned use in the randomized lesion(s) of a bare metal stent (BMS), bioresorbable scaffold (BRS), or non-stent treatment only;
  5. The investigator believes that based on the angiographic appearance that 1) it is unlikely that an OCT catheter can be delivered; 2) if randomized to no IVL, it is unlikely that the lesion(s) can be crossed and pre-dilated by balloon angioplasty alone; 3) if randomized to IVL, it is unlikely that the IVL catheter can be delivered to the lesion (note: pre-dilatation is allowed if necessary for IVL delivery);
  6. Subject has undergone a prior transcatheter or surgical intervention for a non-coronary cardiac condition (e.g. a TAVR or left atrial appendage occlusion) within the prior 6 months, or is anticipated to need such a procedure within 1 year;
  7. Subject has severe stenosis or regurgitation of any heart valve, or moderate aortic stenosis or regurgitation;
  8. Subject has evidence of heart failure by at least one of the following:

  <!-- -->

  1. Left ventricular ejection fraction (LVEF) ≤30% within 1 month prior to enrollment, or
  2. Current heart failure defined as dyspnea with minimal exertion or at rest (NYHA class III or IV within 1 month of the procedure), or
  3. Killip class ≥2 for post STEMI patients; 9.Subject is hemodynamically unstable as evidenced by a SBP of >160 mmHg or <90 mmHg or a heart rate of <50 bpm or >100 bpm (>110 bpm if in atrial fibrillation) 10.Subjects with known allergy to heparin unless bivalirudin will be used as the procedural anticoagulant; 11.Subjects with known allergy to contrast media that cannot be effectively pre-medicated or any prior anaphylaxis to contrast; 12.Subjects with known allergy to aspirin or both clopidogrel and ticagrelor; 13.History of a stroke within 6 months prior to enrollment, excluding transient ischemic attack (TIA) or any prior intracranial bleed; 14.History of active peptic ulcer or upper gastrointestinal bleeding within 6 months prior to enrollment; 15.Inability to tolerate dual antiplatelet therapy for at least 6 months; 16.Known malignancy or any condition with a life expectancy of ≤12 months; 17.Chronic kidney disease (CKD) with an estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m² or on dialysis; 18.Subject has a history of any cognitive or mental health condition that may interfere with the trial participation including all follow-up visits; 19.Subject is a female who is pregnant (women of child-bearing potential must have a negative pregnancy test within 15 days before the procedure); 20.Subject is participating in or has plans to participate in any other investigational drug or device trial that has not reached its primary endpoint.
* Angiographic Exclusion Criteria:

  1. There are no lesions in any target vessel (main epicardial coronary artery including its side branches) that requires treatment that do not meet all angiographic inclusion criteria;
  2. A target lesion is an unprotected LM lesion or an ostial lesion (RCA within 3 mm of the aorta proximal LAD or LCX within 3 mm of the LM);
  3. A target lesion is a true bifurcation with a severely calcified side branch that requires treatment but cannot be treated with IVL because of its size, angulation or other condition. A severely calcified side branch is defined via angiogram as fluoroscopic radiopacities noted without cardiac motion before contrast injection involving both sides of the arterial wall) Note: If a true bifurcation target lesion is included, the main branch must be severely calcified; the side branch may or may not be severely calcified. However, if the side branch is severely calcified, it must be eligible for IVL treatment. Otherwise, the final treatment for the side branch may be balloon angioplasty, a DCB or a DES as per the judgement of the operator. The main branch must be treated with a DES.
  4. A target lesion is totally occluded (100% diameter stenosis with TIMI flow ≤1);
  5. A target lesion contains giant thrombus (defined as angiographic length >2x the reference vessel diameter);
  6. Presence of an aneurysm within 10 mm of the target lesion;
  7. Angiographic evidence of severe dissection (type D - F defined by NHLBI classification) in the target lesion prior to device treatment;
  8. A target vessel has severe or excessive tortuosity or is deemed unsuitable for angioplasty by investigator judgement; Any intent to perform intravascular imaging during the randomization procedure (unless randomized to OCT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3060 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2030-01-20 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) at 3 years | 3 years
  Composite time-to-first event rate of cardiac death, target vessel myocardial infarction (TV-MI), or ischemia-driven target vessel revascularization (iTVR) at 3 years, assessed when the last enrolled patient reaches 1-year follow-up

SECONDARY OUTCOMES:
TVF (at 1 and 2 years) | 1 and 2 years
Target Lesion Failure (TLF) | 30 days, 6 months ,1 year, 2 years, and 3 years
  defined as composite of cardiac death, TVMI, or ischemia-driven target lesion revascularization (iTLR); 3.Major Adverse Cardiovascular Events (MACE), defined as cardiac death, all MI, or TVR;
Major Adverse Cardiovascular Events (MACE) | 30 days, 6 months,1 year, 2 years, and 3 years
  defined as cardiac death, all MI, or TVR;
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 30 days, 6 months,1 year, 2 years, and 3 years
  including all-cause death, MI, stroke, or any revascularization;
Cardiac death | 30 days, 6 months,1 year, 2 years, and 3 years
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all cardiac procedure related deaths including those related to concomitant treatment.
Incidence of stent thrombosis | 30 days, 6 months,1 year, 2 years, and 3 years
  definite or probable stent thrombosis according to the Academic Research Consortium (ARC) criteria.
Severe angiographic complications | Immediate post-procedure
  including type D-F dissection (NHLBI classification), vascular perforation, acute vessel occlusion, persistent slow flow or persistent no-reflow during the procedure;
Procedural strategy success | Immediate post-procedure
  defined as successful passage of the randomized study device through the target lesion, successful study device balloon expansion, successful stent placement with residual stenosis ≤20%, and no occurrence of MACE during hospitalization; Note: Small balloons for pre-dilatation are permitted in the IVL arm. Crossovers to any device (rotational atherectomy, orbital atherectomy, excimer laser, high-pressure, or cutting/scoring balloons) in the IVL arm are defined as a failure. Crossovers to IVL in the BA arm are not permitted but if used (protocol violation), this is a procedural failure. If rotational atherectomy, orbital atherectomy, or excimer laser are required for study device delivery in BA arm, this is also defined as a procedural failure.
Post-procedural minimum stent area (MSA) at the site of maximum calcification and across the entire target lesion; | Immediate post-procedure
Post-procedural mean stent area | Immediate post-procedure
Post-procedural minimum lumen diameter (MLD) | Immediate post-procedure
  MLD refers to the minimum lumen diameter within the stent post-procedure.
Minimum stent expansion | Immediate post-procedure
  Minimum stent expansion is the minimum lumen area within the stent divided by the average of proximal and distal reference lumen areas x 100
Stent malposition | Immediate post-procedure
  defined as distance from stent struts to the vessel wall ≥0.4 mm and the length of stent malposition ≥1 mm;
Number of calcification fractures | Immediate post-procedure
Major and minor edge dissection | Immediate post-procedure
  Edge dissection is classified as major if it involves ≥60 degrees of the vessel circumference at the dissection site and measures ≥3 mm in length or as minor if there is any visible edge dissection involving <60 degrees of the vessel circumference or <3 mm in length;
Major and minor tissue protrusion | Immediate post-procedure
  Tissue protrusion is classified as major if the protrusion area/stent area at the site of tissue protrusion is ≥10% and the minimal intrastent flow area is <90% of the proximal or distal reference area. Note, the minimum in-stent flow area is the minimum value compared with the difference between the stent area and the prolapse area. Tissue protrusion is classified as minor if the protrusion area/stent area at the site of tissue protrusion is <10%, or is ≥10% but the minimal intraluminal flow area is ≥90% of proximal or distal reference area;
Incidence of Untreated reference segment disease | Immediate post-procedure
  Untreated reference segment disease is defined as focal disease with an untreated minimal lumen area (MLA) <4.5 mm2 within 5 mm from the proximal and/or distal stent edges.
Target vessel myocardial infarction (TV-MI) | 30 days, 6 months,1 year, 2 years, and 3 years
  consists of periprocedural MI and spontaneous MI that arise from the target vessel., spontaneous MI using the 4th UDMI, peri-procedural MI using SCAI
ischemia-driven target vessel revascularization (iTVR) | 30 days, 6 months,1 year, 2 years, and 3 years
  repeat revascularization of the target vessel with ischemic symptoms and angiographic evidence
MI | 30 days, 6 months,1 year, 2 years, and 3 years
  consists of periprocedural MI and spontaneous MI, spontaneous MI using the 4th UDMI, peri-procedural MI using SCAI target vessel revascularization, Repeat revascularization of the target vessel
all-cause death | 30 days, 6 months,1 year, 2 years, and 3 years
Stoke | 30 days, 6 months,1 year, 2 years, and 3 years
any revascularization | 30 days, 6 months,1 year, 2 years, and 3 years
Post-procedural mean lumen diameter(LD) | Immediate post-procedure
  LD refers to the average value of lumen diameter measurements calculated by averaging data from all cross-sections throughout the stent
Mean stent expansion | Immediate post-procedure
  Mean stent expansion is the mean stent area (stent volume/analysed stent length) divided by the average of proximal and distal reference lumen areas x 100
Thickness (full-layer or partial) of calcification （mm) | Immediate post-procedure
Depth of calcification fractures(mm） | Immediate post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Principal Investigator — The General Hospital of Northern Theater Command; Gregg W. Stone, Study Chair — Icahn School of Medicine at Mount Sinai, USA
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
This study has no plan to share de-identified individual participant data (IPD) with researchers outside the primary study team. The reasons for this decision are as follows:
  Informed Consent & Ethical Commitment: The informed consent documents for this study do not include provisions for IPD sharing, as participants only consented to data use for the original analysis of this study. This approach has been reviewed and approved by the Institutional Review Board/Ethics Committee (IRB/IEC) to uphold ethical commitments and avoid using data beyond the scope of participant understanding.

REFERENCES:
- [Result] [16] Han Y, Jing Q, Liu H, et al. A novel coronary intravascular Lithotripsy device in patients with severely calcified lesions: LEAD-FIM study. Presented at EuroPCR 2024.
- [Result] [15] Kirtane AJ, Généreux P, Lewis B, Shlofmitz RA, Dohad S, Choudary J, Dahle T, Pineda AM, Shunk K, Maehara A, Popma A, Redfors B, Ali ZA, Krucoff M, Armstrong E, Kandzari DE, O'Neill W, Kraemer C, Stiefel KM, Jones DE, Chambers J, Stone GW; ECLIPSE Investigators. Orbital atherectomy versus balloon angioplasty before drug-eluting stent implantation in severely calcified lesions eligible for both treatment strategies (ECLIPSE): a multicentre, open-label, randomised trial. Lancet. 2025 Apr 12;405(10486):1240-1251.
- [Result] [14] Moussa ID, Klein LW, Shah B et al. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Journal Pre-proof Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013; 62:1563-70
- [Result] [13] Blachutzik F, Meier S, Weissner M, et al. Comparison of coronary intravascular lithotripsy and rotational atherectomy in the modification of severely calcified stenosis[J]. Am J Cardiol,2023,197: 93-100. DOI: 10.1016/j.amjcard.2023.02.028.
- [Result] [12] Mousa MAA, Bingen BO, Al Amri I, et al. Efficacy and safety of intravascular lithotripsy versus rotational atherectomy in balloon-crossable heavily calcified coronary lesions [J]. Cardiovasc Revasc Med, 2023,48: 1-6.
- [Result] [11] Cubero-Gallego H, Calvo-Fernandez A, Tizon-Marcos H, et al. Real-world multicenter coronary lithotripsy registry: long-term clinical follow-up[J]. J Invasive Cardiol, 2022, 34(10)：E701-E708.
- [Result] [10] Wong B， El-Jack S， Newcombe R， et al. Shockwave intravascular lithotripsy for calcified coronary lesions： first real-world experience[J]. J Invasive Cardiol, 2019, 31(3):46-48.
- [Result] [9] Rodriguez-Leor, O, Cid-Alvarez, A, Lopez-Benito, M. et al. A Prospective, Multicenter, Real-World Registry of Coronary Lithotripsy in Calcified Coronary Arteries: The REPLICA-EPIC18 Study. J Am Coll Cardiol Intv. 2024 Mar, 17 (6) 756-767.
- [Result] [8] Tian F， Zhou SS， Liu JH， et al. Treatment of severely calcified coronary artery disease by intravascular lithotripsy primary outcomes and 180-day follow-up from the Chinese SOLSTICE Trial [J]. J Geriatr Cardiol， 2023, 20(1)： 32-39. DOI：10.26599/1671-5411.2023.01.005.
- [Result] [7] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646.
- [Result] [6] Saito S, Yamazaki S, Takahashi A, et al. Intravascular Lithotripsy for Vessel Preparation in Severely Calcified Coronary Arteries Prior to Stent Placement - Primary Outcomes from the Japanese Disrupt CAD IV Study. Circ J.2021 May 25;85(6):826-833.
- [Result] Kereiakes DJ, Hill JM, Ben-Yehuda O, Maehara A, Alexander B, Stone GW. Evaluation of safety and efficacy of coronary intravascular lithotripsy for treatment of severely calcified coronary stenoses: Design and rationale for the Disrupt CAD III trial. Am Heart J. 2020 Jul; 225:10-18. doi: 10.1016/j.ahj.2020.04.005.
- [Result] Hill JM, Kereiakes DJ, et al. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603.
- [Result] Ali ZA, Nef H, et al. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10): e008434.
- [Result] Brinton TJ, et al. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836.
- [Result] Chinese Society of Cardiology, Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. Guidelines for percutaneous coronary intervention (2025). Zhonghua Xin Xue Guan Bing Za Zhi. 2025 Jun 12; 53:16-44. Chinese. doi: 10.3760/cma.j.cn112148-20250422-00302. Epub ahead of print.